CLINICAL TRIAL: NCT00320554
Title: Motion Characteristics of the Foot and Ankle as Measured by Durometer Readings
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Other Study IDs: SR040406008
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Foot Motion Characteristics

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Durometer analysis

SUMMARY:
The purpose of this study is to determine the motion characteristics of the foot and ankle with a durometer as a method of measurement.

DETAILED DESCRIPTION:
This study will assess and establish the motion characteristics of the foot and ankle with the use of a durometer as a measure of motion patterns.

The durometer is a device commonly used in materials testing that measures displacement through the use of a piezoelectric sensor configured to detect motion a in the form of a reflected wave back from the surface being tested.

ELIGIBILITY:
Inclusion Criteria: Logan student, staff, or faculty with no history of ankle injury; 2. Age 18 - 60 yoa Exclusion Criteria: 1. Logan student, staff, or faculty with no history of ankle surgery 1. No visual or vestibular condition that would affect balance; 2. Systemic illness that have an adverse effect on balance; 3. Local infection, injury or other malignancy affecting the lower extremity; 4. Any unstable joints of the lower extremity; 5. Any manipulation to the foot ankle joints within 48 hours; 6. Prescription or herbal muscle stimulants, relaxants, etc.; 7. Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Enix, DC, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States